CLINICAL TRIAL: NCT03585023
Title: Silent Intracellular Infections and Early Pregnancy Loss
Brief Title: Infections and Pregnancy Loss: Correlation Between Abortion and Silent Infections.
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Angela Graziano, Doctor, University Hospital of Ferrara
Other Study IDs: PRUA1GR-2013-00000220
Record Dates: First submitted 2018-06-04; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Pregnancy Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All samples, both spontaneous (spontaneous miscarriage) and elective (voluntary interruption of pregnancy), will be obtained after uterine cavity curettage.
  All women underwent PBMC extraction from peripheral whole blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spontaneous miscarriage: The study group will be recruited at admission for uterine cavity revision planned for spontaneous abortion.
  Interventions: Diagnostic Test: Spontaneous miscarriage; Diagnostic Test: Voluntary pregnancy interruption
- Voluntary pregnancy interruption: The control group will be recruited at admission for uterine cavity revision planned for voluntary pregnancy interruption.
  Interventions: Diagnostic Test: Spontaneous miscarriage; Diagnostic Test: Voluntary pregnancy interruption

INTERVENTIONS:
Diagnostic Test: Spontaneous miscarriage — Viral DNA and RNA analysis of HPyV and HPV, BKV and JCV. Bacterial DNA and RNA analysis of Chlamydia trachomatis, Ureaplasma parvum, U. urealyticum, Mycoplasma hominis.
Diagnostic Test: Voluntary pregnancy interruption — Viral DNA and RNA analysis of HPyV and HPV, BKV and JCV. Bacterial DNA and RNA analysis of Chlamydia trachomatis, Ureaplasma parvum, U. urealyticum, Mycoplasma hominis.

SUMMARY:
Correlation between the presence of intracellular viruses/bacteria and the incidence of miscarriage during the first trimester of pregnancy.

DETAILED DESCRIPTION:
In this study we will analyse chorionic villi derived from abortion during the first trimester of pregnancy (spontaneous abortion vs voluntary pregnancy interruption), in order to correlate the presence of infective viruses/bacteria and the incidence of miscarriage.

The first objective of this project will be to find the viral DNA of HPV, BK and JC polyomaviruses and bacterial DNA of Chlamydia trachomatis, Ureaplasma parvum, Ureaplasma urealyticum, Mycoplasma hominis in the aborted tissues collected from spontaneous abortions, and to compare the prevalence of these DNAs to those derived from elective specimens.

Acronyms:

DNA: deoxyribonucleic acid HPV: human papillomavirus PCR: polymerase chain reaction HPyV: human polyomavirus PBMC: peripheral blood mononucleated cell BKV: BK polyomavirus JCV: JC polyomavirus

ELIGIBILITY:
I.Inclusion and exclusion criteria

Inclusion criteria:

* age of the patients range from 18 to 42 years old;
* gestational age ranging in the first 12 weeks.

Exclusion criteria:

* medical history or laboratory tests positive for sexually transmitted diseases (HIV, HBV, HCV, LUE) during the last year;
* Congenital or Acquired Immunodeficiency diseases, or immunosuppressive therapies during the last year;
* Therapeutic abortion (voluntary interruption of pregnancy, law 194 art 6 comma b)
* well known causes responsable for spontaneous abortions such as genetic, severe uterine or hormonal abnormalities and use of teratogenic drugs.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women
Study Population: Women who underwent revision of uterine cavity for spontaneous abortion or voluntary termination of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-11-15 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2017-05-14 (Actual)

PRIMARY OUTCOMES:
Individuation of DNA of intracellular agents (viral und bacterial) in chorionic tissue und blood sample. | December 2014 - April 2017
  The primary outcome of this project is to find the DNA of viral (HPV, HPyV,BK and JC), or bacterial agents (Chlamydia trachomatis, Ureaplasma parvum, U. urealyticum, Mycoplasma hominis) in samples obtained from spontaneous abortion or elective interruption of pregnancy.